CLINICAL TRIAL: NCT05921539
Title: Does Axillary Nerve and Inferior Capsule Release Add Extra Benefit to Steroid Hydrodilatation in Treating Patients With Adhesive Capsulitis
Brief Title: Does Axillary Nerve and Inferior Capsule Release Add Extra Benefit in Treating Patients With Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-02-011B
Record Dates: First submitted 2021-11-22; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-01

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrodilatation and axillary nerve injection (Experimental): patient received ultrasound-guided steroid hydrodilatation via posterior recess
  Interventions: Drug: steroid hydrodilatation; Drug: axillary nerve injection
- hydrodilatation only (Active Comparator): patient received ultrasound-guided steroid hydrodilatation only
  Interventions: Drug: steroid hydrodilatation

INTERVENTIONS:
Drug: steroid hydrodilatation — ultrasound-guided steroid hydrodilatation
Drug: axillary nerve injection — ultrasound-guided axillary nerve injection
  Arms: hydrodilatation and axillary nerve injection

SUMMARY:
This study was conducted to compare the efficacy of hydrodilatation with steroid via posterior approach versus hydrodilatation with steroid with axillary nerve injection for treating patients with adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis is a common cause of shoulder pain, and the efficacy of most interventions is limited. This study was conducted to compare the efficacy of rotator interval injection with steroid with that of steroid hydrodilatatoin for treating adhesive capsulitis.

Design: a prospective, single-blinded, randomized, clinical trial

Patient and methods:

Patients with adhesive capsulitis were enrolled and randomly allocated into group 1 ( ultrasound guided hydrodilatation with steroid via posterior approach) and group 2 (ultrasound guided hydrodilatation with steroid via posterior approach as well as axillary nerve injection). The patients were evaluated before treatment and were reevaluated 0, 6, and 12 weeks after the beginning of the treatment. Outcomes measures included a pain scale (visual analog scale), range of motion, and Shoulder Pain And Disability Index.

ELIGIBILITY:
Inclusion Criteria:

1. age 35-65 years (to prevent the inclusion of patients with secondary AC),
2. onset of shoulder stiffness since over a month
3. limitation in the passive range of motion (ROM) over 30° when compared with the contralateral side in at least two of these three movements: forward flexion, abduction, or external rotation.

Exclusion Criteria:

1. ultrasound findings of rotator cuff tears
2. plain radiography findings of significant glenohumeral joint arthritis
3. accompanying cervical radiculopathy
4. systemic inflammatory joint disease
5. intra-articular injection into the glenohumeral joint within the past 3 months
6. history of surgery on the affected shoulders
7. regular use of systemic non-steroidal anti-inflammatory drugs or corticosteroids
8. allergy to corticosteroid or lidocaine. -

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain And disability index | Change of the score between 6 weeks and baseline, and change of the score between 12 weeks and baseline
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.function. The score is divided into four sections: pain, activity of daily living, ROM and strength

SECONDARY OUTCOMES:
pain intensity | Change of the score between 6 weeks and baseline, and change of the score between 12 weeks and baseline
  pain intensity was measured by visual analog scale. Each patient was asked to indicate his/her current level of pain by marking a point on a 100-mm VAS, for which 0 represented no pain and 100 represented unbearable pain.
glenohumeral joint range of motion | Change at baseline, 6 weeks, 12 weeks
  change in degrees of shoulder motion

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No